CLINICAL TRIAL: NCT00484432
Title: NGR012: A Phase II Study of NGR-hTNF Administered in Combination With Doxorubicin Every 3 Weeks in Patients Affected by Advanced or Metastatic Ovarian Cancer
Brief Title: Study of NGR-hTNF in Combination With Doxorubicin in Patients Affected by Advanced or Metastatic Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGR012; 2007-000004-33 (EudraCT Number)
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Ovarian Cancer Metastatic Recurrent
Keywords: NGR-hTNF; Ovarian cancer; Doxorubicin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A: NGR-hTNF + doxorubicin (Experimental): NGR-hTNF plus doxorubicin
  Interventions: Drug: NGR-hTNF; Drug: doxorubicin

INTERVENTIONS:
Drug: NGR-hTNF — NGR-hTNF: 0.8 mcg/m² as 60-minute intravenous infusion every 3 week until confirmed evidence of disease progression or unacceptable toxicity occurs
Drug: doxorubicin — Doxorubicin: 60mg/m² every 3 weeks, until cumulative dose of 550 mg/m²

SUMMARY:
The main objective of the trial is to document the response rate in patients affected by metastatic ovarian cancer, treated with NGR-hTNF plus doxorubicin. Safety will be established by clinical and laboratory assessment according to NCI-CTC criteria.

DETAILED DESCRIPTION:
This is a phase II, open-label,single arm, non-randomized study that will be conducted in patients affected by metastatic ovarian cancer, that will be conducted using Simon's two-stage design method.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old affected by advanced or metastatic ovarian cancer previously treated with platinum regimens (cis or carboplatin) plus paclitaxel and with documented progression disease within 6 months from last chemotherapy administered (refractory/resistant population) or in progression disease after 6 months from last chemotherapy (platinum regimens plus paclitaxel) administered
* Rechallenge with platinum regimens
* No previous exposure to anthracyclines
* Histologically or cytologically confirmed ovarian carcinoma
* Life expectancy more than 3 months
* ECOG Performance status 0 - 1
* Normal cardiac function (LVEF ≥55%) and absence of uncontrolled hypertension
* Measurable disease defined as ≥1 unidimensional measurable lesion ≥ 20 mm by conventional technics or ≥ 10 mm ( spiral CT scan or PET); ascites is allowed if present with peritoneal carcinosis
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

  * Neutrophils > 1.5 x 10^9/L and platelets > 100 x 10^9/L
  * Bilirubin < 1.5 x ULN
  * AST and/or ALT < 2.5 x ULN in absence of liver metastasis
  * AST and/or ALT < 5 x ULN in presence of liver metastasis
  * Serum creatinine < 1.5 x ULN
* Patients may have had prior therapy providing the following conditions are met:

  * Chemotherapy and radiotherapy: wash-out period of 28 days
  * Surgery: wash-out period of 14 days
* Absence of any conditions in which hypervolaemia and its consequences (e.g. increased stroke volume, elevated blood pressure) or haemodilution could represent a risk for the patient (take as reference "Technical data sheet human albumin" specifically used in Pharmacy Department for NGR-hTNF dilution)
* Patients must give written informed consent to participate in the study

Exclusion criteria:

* Concurrent anticancer therapy
* Patients must not receive any other investigational agents while on study
* New York Heart Association class II-IV cardiac disease
* Acute angina
* Patients with myocardial infarction within the last six (6) months
* Patient with significant peripheral vascular disease
* Thrombosis of main portal vein
* Clinical signs of CNS involvement
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Antitumor activity defined as response rate | during the study
  Evaluated according to Response evaluation criteria in solid tumors (RECIST)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | during the study
  PFS evaluated according to Response evaluation criteria in solid tumors (RECIST)
Overall survival (OS) | from the date of randomization to the date of death, assessed up to 6 months
  Defined as the time from the date of randomization until the date of death due to any cause or the last date the patient was known to be alive
CA125 (U/mL) measurement | from the randomization, every 6 weeks until the end of treatment
  Tumor marker evaluation
Safety according to NCI-CTCAE criteria (version 3) | during the study
  To evaluate safety profile related to NGR-hTNF

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (2):
- Italy (2):
  - Fondazione San Raffaele del Monte Tabor, Milan
  - Policlinico Universitario A. Gemelli, Rome

REFERENCES:
- [Result] Lorusso D, Scambia G, Amadio G, di Legge A, Pietragalla A, De Vincenzo R, Masciullo V, Di Stefano M, Mangili G, Citterio G, Mantori M, Lambiase A, Bordignon C. Phase II study of NGR-hTNF in combination with doxorubicin in relapsed ovarian cancer patients. Br J Cancer. 2012 Jun 26;107(1):37-42. doi: 10.1038/bjc.2012.233. Epub 2012 May 29. PMID 22644293